CLINICAL TRIAL: NCT06350981
Title: Analgesic Requirement for Post-Operative Pain Control in Elective 1-3 Level Transforaminal Lumbar Interbody Fusion: Comparison of Thoracolumbar Interfascial Plane Block With Exparel to Bupivacaine HCl
Brief Title: Analgesic Requirement for Post-Operative Pain Control in TLIP Interbody Fusion
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FORE813
Record Dates: First submitted 2024-03-15; First posted 2024-04-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Back Pain; Surgery-Complications; Narcotic Use; Physical Stress; Post Operative Pain
MeSH Terms: conditions — Back Pain; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study subjects will be randomized to either Group 1 or Group 2 in a 1:1 ratio based on the randomization scheme in sealed envelopes maintained by the study coordinator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel TLIP Injection (Experimental): Subjects will receive 20 mL of EXPAREL 266mg mixed with 10 mL of 0.25% bupivacaine. A total of 30 mL of mixed solution is injected into the thoracolumbar interfacial plane.
  Interventions: Drug: Exparel
- Bupivicaine HCL TLIP Injection (Active Comparator): Standard of care will consist of 0.25% Bupivacaine HCl TLIP injection. Subjects will receive 30 mL of the solution, injected into the thoracolumbar interfacial plane.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Exparel — 20 mL of EXPAREL 266mg mixed with 10 mL of 0.25% bupivacaine
  Arms: Exparel TLIP Injection
Drug: Bupivacain — Standard of care will consist of 0.25% Bupivacaine HCl TLIP injection 30mL
  Arms: Bupivicaine HCL TLIP Injection

SUMMARY:
The goal of this clinical trail is to to compare the efficacy of thoracolumbar interfascial plane block with Exparel vs with standard of care 0.25% Bupivacaine HCl in patients undergoing 1-3 level elective transforaminal lumbar interbody fusion. The investigators hypothesize that thoracolumbar interfascial plane block with Exparel will outperform standard of care (supplemented with interfascial plane block of 0.25% Bupivacaine HCl) with regards to pain reduction, narcotic use, length of hospital stay, time to mobilization with physical therapy, narcotic usage in the hospital, and post operative pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older,
* Patients admitted to AHC for 1-3 level TLIF,
* Patients who have given written informed consent,
* BMI between 18-35 kg/m2,

Exclusion Criteria:

* Patients with known allergic reactions to standard of care analgesics,
* Female patients who are pregnant
* Patients with any previous lumbar spine instrumented surgery,
* Chronic opioid use within 30 days prior to randomization that exceeds average ≥30 oral morphine equivalents/day,
* Patients with known allergy to local anesthetics,
* Patients with known or suspected to have neuromuscular disorders impairing neuromuscular blockade (e.g. myasthenia gravis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Compare efficacy of thoracolumbar interfacial plane block with Exparel vs. standard of care (0.25% Bupivacaine HCL) is surgical subjects undergoing 1-3 level elective transforaminal lumbar interbody fusion. | 0-72 hours post-operatively
  Data will be analyzed by randomized treatment group to determine efficacy. Superiority of treatment with EXPAREL compared with Bupivacaine hydrochloride will be determined using linear regression adjusting for Pain Catastrophizing Scale with treatment as main effect for the primary efficacy endpoint of area under the curve of the Numerical rating scale pain intensity scores from 0 to 72 hours post-surgery.

SECONDARY OUTCOMES:
Total Postsurgical opioid consumption | 0-72 hours postoperatively
  The following data points will be recorded to further claim the investigators hypothesis of treatment with EXPAREL compared to Bupivacaine hydrochloride.
  • Total postsurgical opioid consumption in oral morphine equivalents (Oral morphine equivalents) from 0 to 76 hours post-surgery
Time to discharge | 0-72 hours postoperatively
  collect hours of hospital stay
Time to ambulation | 0-72 hours postoperatively
  collect time ambulated from surgery
Maximum ambulated distance | 0-72 hours postoperatively
  Physical Therapy will document the distance subject could ambulate after surgery
Numeric Rating Pain Scale (Physical Therapy) | 0-72 hours postoperatively
  Measure pain score (scale of 0-10 with 0 indicates no pain and 10 severe pain) during physical therapy (ambulation)
Numeric Rating Pain Scale | 0-72 hours with additional follow-up at 14 days (first clinic visit)
  Numerical rating scale pain intensity scores at 24hour, 36hour, 60hour, and 72hour from the end of surgery and again at the first clinic visit postoperatively (scale of 0-10 with 0 indicates no pain and 10 severe pain)
Oswestry Disability Index (ODI) | 0- 14 days postoperatively
  10 questions relating to function specific to low back pain given before surgery and collected at 14 day post op visit.
Pain Catastrophizing Scale (PCS) | 0-14 days postoperatively
  This scale measures thoughts and feelings that may be associated with pain. it is rated 0-5 with 0 indicating not at all, 1 indicating to a slight degree, 2 indicates a moderate degree, 3 indicates a great degree and 4 idicates all the time.
  There are 13 statements that are rated, the ratings are scored to determine where each subject falls in the scale.

CONTACTS AND LOCATIONS:
Overall Officials: John Small, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Foundation for Orthopaedic Research and Education, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No